CLINICAL TRIAL: NCT07283926
Title: Tailored Medical Nutrition Therapy Meal Delivery for the Vulnerable Food Insecure Elderly Patients With End Stage Kidney Disease on Haemodialysis: A Feasibility Pilot Study
Brief Title: Restorative and Supportive Meals at HomeCare
Acronym: RASA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Wai Yew Yang, Senior Lecturer, Universiti Putra Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: JKEUPM-2025-321; VOT 6300570 (Other Grant/Funding Number: Pak Rashid Foundation (Yayasan Pak Rashid))
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease on Hemodialysis; Meals; Medical Nutrition Therapy
Keywords: medical nutrition therapy; meal delivery; hemodialysis; elderly; food security; socioeconomic
MeSH Terms: interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: This study is designed as a sequential single arm crossover intervention study of phase 1 (menu design and cost analysis) and phase 2 (intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Sequential single arm crossover intervention study:
  1. Phase 1 (menu design and cost analysis)
     * Menu planning for tailored MNT diet suitable for elderly patients with chronic kidney disease on hemodialysis
     * Pilot testing of newly developed menu including sensory evaluation
     * Finalise standard recipes including nutrients, cost and hygiene analysis
  2. Phase 2 (intervention)
  a) Participant's enrolment Interested participants will undergo screening and selection based on the inclusion criteria and exclusion criteria b) Time-point and Data collection Participants will undergo testing at each time-point of baseline (0 month), after 4 weeks (1 month), and 8 weeks (2 month): food insecurity tool, malnutrition assessment tool, body composition assessment, clinical assessment and dietary assessment c) Participants will provide satisfaction assessment (SERQUAL questionnaire) d) Participants will follow usual diet for 4 weeks (control period), followed by 4 weeks on the MNT meals
  Interventions: Other: Medical Nutrition Therapy + Meal Delivery

INTERVENTIONS:
Other: Medical Nutrition Therapy + Meal Delivery — The tailored medical nutrition therapy menu is planned to meet the requirement of elderly chronic kidney disease patients on hemodialysis following the needs assessment on their existing nutritional status. The menu planning is completed by registered dietitians, and the vegetables are planted and supplied by certified agriculturist adhering to the local farming standards. The recipes are analysed with the nutrients, cost and hygiene to ensure its practicality, accessibility, affordability and safety.
  Other Names: RASA (Restorative And Supportive Meals At HomeCare)

SUMMARY:
The pilot intervention study is designed to evaluate the feasibility of implementing a tailored medical nutrition therapy (MNT) meal-delivery for 25 elderly, low-income food insecure patients with end-stage kidney disease undergoing maintenance hemodialysis at dialysis centers. Following comprehensive baseline assessments, participants will first maintain their usual dietary patterns for a 4-week control period to establish baseline nutritional and clinical parameters. This will be followed by a 4-week intervention period during which participants will receive individually tailored MNT meals designed to meet their renal-specific nutritional requirements, including energy, protein, potassium, phosphate and sodium intake. Weekly monitoring during dialysis sessions will include assessment of adherence, dietary intake, and clinical tolerance, providing detailed insights into the feasibility, safety, and potential clinical impact of the tailored nutrition intervention in this vulnerable population.

DETAILED DESCRIPTION:
Background Malaysia is expecting population ageing with a projection of 15% of Malaysia's population will be over 65 years by 2030. Older adults often face challenges related to food insecurity and chronic disease management, which affect their overall well-being. In 2018, 10.4% of older adults were classified as food insecure, and this number is projected to escalate with the growing older adult population. On the other hand, those suffering from chronic kidney disease (CKD) face one of the most difficult diets among clinical patients. With economic constraints, the elderly's abilities to acquire the right food could be limited, predisposing them to increased morbidity and mortality. While much work is needed to ascertain the complex interplay between food insecurity, chronic disease management, and well-being in this population, a tailored intervention programme could help improve food security and health status, yet it is not well researched.

Problem Statement Food insecure elderly patients with end-stage renal disease (ESRD) on haemodialysis (HD) in Malaysia have low adherence on renal diet and are at the highest risk of malnutrition and food-borne illness predisposing them to increased morbidity and mortality.

Justification of Study At present, there is limited evidence on availability of a tailored medical nutrition therapy (MNT) meal delivery specific for HD patients in Malaysia. While much work is needed to ascertain the complex interplay between food insecurity, chronic disease management, and well-being, a tailored intervention programme could help improve the food security and health status of elderly population in Malaysia.

Research Question(s) Can tailored MNT meal delivery improve food safety, food insecurity and nutritional status of food insecure malnourished elderly patients with ESRD on HD?

Research objectives

General Objective:

To determine the feasibility of tailored medical nutrition therapy meal delivery intervention programme for elderly patients undergoing haemodialysis

Specific Objectives:

To examine the effectiveness of tailored MNT meal delivery on food safety, food insecurity and nutritional status of food insecure elderly patients with end stage kidney disease on haemodialysis

Research methodology To accomplish the objective, a single arm crossover study is proposed to be conducted over a one-year period divided into two phases: Phase One (menu planning) and Phase Two (intervention) among food insecure malnourished elderly patients on haemodialysis. Data will be collected at 3-time points on food insecurity, nutritional status and meal satisfaction.

Expected outcomes

1. Potentially improve nutritional intake among food insecure elderly patients on haemodialysis by using self-grown vegetables that follows good practices in Malaysian Good Agricultural Practices with good handling of post-harvest management;
2. Extend the understanding of interplay between food insecurity, chronic disease management, and well-being of older adults, and;
3. Establish link between community, university and industry on affordable, tailored therapeutic meals for vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with chronic kidney disease on hemodialysis aged 60 and above (receiving hemodialysis treatment ≥3 days/week, dialysis vintage ≥3 months), and received at least one nutrition consultation by dietitian;
* From the low-income households based on the Malaysia's Department of Statistics criteria and food insecure;
* With co-morbidities of hypertension and cardiovascular disease;
* Consent to participate for 2 months period

Exclusion Criteria:

* Patients with chronic kidney disease on hemodialysis aged 59 and below, patients undergoing peritoneal dialysis/alternate hemodialysis and peritoneal dialysis/ dialysis vintage <3 months), and have not received at least one nutrition consultation by dietitian;
* From non low-income households based on the Malaysia's Department of Statistics criteria and food insecure
* With co-morbidities aside from those mentioned above (i.e. diabetes, cancer, gastrointestinal disorders, liver disease or any chronic diseases requiring specialised medical nutrition therapy)
* Patients diagnosed with food allergies or intolerance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | From enrollment to the end of intervention at 8 weeks
  The nutritional status of hemodialysis patients is assessed based on the presence of protein-energy wasting (PEW), categorised as either "yes" or "no." PEW is diagnosed according to the diagnostic criteria established by International Society of Renal Nutrition and Metabolism (ISRNM). Four main categories will be evaluated to diagnose PEW: (1) Serum chemistry; (2) Body mass; (3) Muscle mass; and (4) Dietary intake. The subject is diagnosed with PEW if at least three out of these four listed categories are met, with at least one diagnostic test conducted within each category

SECONDARY OUTCOMES:
Blood Profile (Hemoglobin) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Hemoglobin, g/dL) to determine number of participants with abnormal laboratory tests results.
Blood Profile (Albumn) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Albumin g/L) to determine number of participants with abnormal laboratory tests results.
Blood Profile (Sodium) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Sodium - mmol/L) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Potassium) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Potassium - mmol/L) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Phosphate) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Phosphate - mmol/L) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Calcium) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Calcium - mmol/L) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Lipid Profile) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Lipid Profile - mmol/L) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Glycated hemoglobin - HbA1C) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Glycated hemoglobin - HbA1C in percentage) to determine the number of participants with abnormal laboratory tests results
Blood Profile (Total Iron Binding Capacity) | From enrollment to the end of intervention at 8 weeks
  Assessed using standard laboratory methods from routine blood samples collected during dialysis sessions (Total Iron Binding Capacity - umol/L) to determine the number of participants with abnormal laboratory tests results
Anthropometry markers (weight) | From enrollment to the end of intervention at 8 weeks
  The following measurements will be determined on weight in kg (dry weight, pre and post-hemodialysis) for the calculation of body mass index:
  * Dry weight to be obtain from medical record as determined by the nephrologist
  * Pre-Dialysis Weight: Weight to be taken before hemodialysis session
  * Post-Dialysis Weight: Weight to be taken after hemodialysis session
Anthropometry markers (height) | From enrollment to the end of intervention at 8 weeks
  The measurements will be determined on height in metre for the calculation of body mass index
Body Composition (Mid-arm circumference) | From enrollment to the end of intervention at 8 weeks
  Measurements on the following will be performed on mid-arm circumference (MAC) by identifying the midpoint of shoulder and elbow on the non-fistula arm, then wrap the arm with measuring tape to determine number of participants with abnormal body composition results
Body Composition (Triceps skinfold) | From enrollment to the end of intervention at 8 weeks
  Measurements on the following will be performed triceps skinfold by identifying the midpoint of shoulder and elbow on the non-fistula arm, then grasp a vertical skinfold and lift perpendicular, then measure using skinfold calliper to determine number of participants with abnormal body composition results
Body Composition (Body fat percentage) | From enrollment to the end of intervention at 8 weeks
  Measurements on the following will be performed using a bioimpedance equipment (in percentage) to determine number of participants with abnormal body composition results
Body Composition (Skeletal muscle) | From enrollment to the end of intervention at 8 weeks
  Measurements on the following will be performed using a bioimpedance equipment (in cm) to determine number of participants with abnormal body composition results
Food Insecurity (FIES) | From enrollment to the end of intervention at 8 weeks
  Assessed using the Food Insecurity Experience Scale (FIES) through an interview-based questionnaire to evaluate participants' experiences and access to adequate food over the past 12 months. The FIES-SM consists of eight questions with dichotomous yes or no responses. The responses are coded as 1 for "yes", 0 for "no" and N/A for "Don't know" or "Refused". The responses were then summed to yield raw scores ranging from 0 to 8. Responses with raw scores = 0 to 3, will be classified as food secure, raw scores = 4 to 6 will be considered as moderate food insecurity, and raw scores = 7 to 8 will be categorised as severe food insecurity.
Dietary Intake | From enrollment to the end of intervention at 8 weeks
  The dietary energy intake (DEI) and dietary protein intake (DPI) are estimated using a diet history interview for dialysis and non-dialysis day.
  During the intervention phase, participants will be provided with a food diary to record all meals and snacks consumed.
  Nutrient analysis is then calculated from these reports.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Yew Yang, PhD; MMedSci; BSc, Principal Investigator — Universiti Putra Malaysia
Locations (4):
- Malaysia (4):
  - NKF Good Health (Kampung Pandan), Kuala Lumpur, Kuala Lumpur
  - NKF Calvary, Kuala Lumpur, Kuala Lumpur
  - NKF Rotary Damansara (Selayang), Batu Caves, Selangor
  - NKF Charis, Cheras, Wilayah Persekutuan Kuala Lumpu

IPD SHARING:
Plan to Share IPD: Undecided
The privacy and confidentiality of the participants are of concern to be shared in public domain.